CLINICAL TRIAL: NCT05306249
Title: Effects of Cannabidiol (CBD) on the Activation of Autophagy and Inflammation Genes, Functional Consequences in Virologically Controlled HIV-infected Patients
Acronym: GALIG-CBD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHRO-2021-01
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: HIV Seropositivity
Keywords: HIV-1; CBD
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBD LGP 50 group (Experimental): Patients will receive CBD LGP 50 at a dose of 1 mg/kg twice a day in the form of oil dispensed through a graduated pipette until the end of week 12.
  Interventions: Drug: CBD LGP 50
- Control group (Placebo Comparator): Patients will receive the MCT oil placebo without CBD until the end of week 12.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CBD LGP 50 — Patients will receive CBD LGP 50 at a dose of 1 mg/kg twice a day in the form of oil dispensed through a graduated pipette until the end of week 12.
  Arms: CBD LGP 50 group
Drug: Placebo — Patients will receive the MCT oil placebo without CBD until the end of week 12.
  Arms: Control group

SUMMARY:
Autophagy and apoptosis are natural cellular mechanisms which consist for the first in a recycling and elimination process of potentially toxic cellular waste, and for the second in a process of cellular suicide when it becomes abnormal and "not" repairable, notably by autophagy. A deficit in autophagic function at the cellular level can lead to chronic inflammation and accelerated cellular senescence. Apoptosis is a beneficial phenomenon because it eliminates abnormal cells that could endanger the organism if it survives (e.g. karyotypic atypia). Uncontrolled, it can be deleterious if apoptosis is hypo or hyperactive.

DETAILED DESCRIPTION:
The Centre of Molecular Biology of the CNRS in Orléans has developed for many years an expertise concerning apoptosis via the discovery of the GALIG gene. This pro-apoptotic gene produces two proteins, one of which, cytogaligin, interacts with several proteins involved in autophagy.

Recent translational research conducted jointly by the CNRS and CHR Orléans teams have shown that PBMC from HIV-infected patients who have been on effective cART for at least 4 years show changes in the expression of certain genes involved in autophagy (BECN1, GABARAPL1, MAP1LC3B and GALIG). Gomez-Mora et al. also reported a decrease in autophagic function in CD4+ T cells of patients, with the impairment of autophagy being more important as the reconstitution of the CD4+ T compartment is incomplete. Thus, autophagy defects are more pronounced in patients whose CD4 T cell count remains low, suggesting a link between autophagy and CD4 T cell depletion.In summary, even after prolonged virological control and apparent immune reconstitution, PLWH (people living with HIV) exhibit deregulation of genes involved in autophagy.

In the simian model, Δ9-tetrahydrocannabinol (Δ9-THC) cannabinoids would reduce inflammation associated with intestinal tissues, but also SIV viral load and mortality in males only. A recent review points to the potential benefit of cannabinoids on inflammation in the context of HIV. PLHIV who regularly use cannabis, and therefore potentially exposed to Δ9-THC and cannabidiol (CBD), have been the subject of a significant literature. Thus, it has been reported that in these patients, compared to non-consumers, there is a greater reduction in the HIV reservoir (HIV-DNA), a decrease in activated monocytes, the latter being linked to inflammation, as well as a reduced activation of CD4+ and CD8+ lymphocytes.

A first analysis is based on 6 HIV+ patients virologically controlled for at least 4 years, having absorbed, as a dietary supplement, for 4 weeks a dose of 30 mg x2 per day of CBD duly controlled pharmacologically (Δ9-THC dosage < 0.1%) and having declared not to use drugs. We were able to note by discriminant factor analysis (DFA):

* a significant change in the expression of genes involved in autophagy. Their activation profile of genes involved in autophagy is no longer identical to that of virologically controlled HIV+ patients who did not take CBD.
* a profile of serum inflammatory cytokines that is close to the profile of HIV-negative individuals, but different from that of PLWHIV who have not consumed CBD.

Thus, CBD, which has no psychotropic effect, could have beneficial effects on HIV patients by reducing cellular senescence, inflammation and their consequences in terms of co-morbidities as well as the level of HIV reservoirs through an apoptotic phenomenon of cells hosting HIV in a quiescent state. Among the molecules present in the plant and in particular the species Cannabis sativa L., can be present the CBD, the Δ9 THC and a multitude of terpenes without psychotropic effects, which would be responsible for an "effect of entourage". Studies argue for a synergistic effect of these molecules to lead to the suspected effects.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient aged 18 or over at the time of signing the informed consent.
* Adults living with HIV1 not co-infected with HIV2
* Documented evidence of HIV plasma RNA assays <50 copies per ml during the 3 years preceding the inclusion, including tolerance of a few occasional "blips",
* HIV 1 plasma RNA assay <50 copies / ml at inclusion
* Patient whose current antiretroviral therapy has not been interrupted during the three months prior to inclusion
* Patient not taking recreational drugs including cannabis in the past six months
* Affiliated with social security
* Men or women. Women must not be pregnant or breastfeeding. If they are of childbearing potential, they should receive active contraception.
* Be able to give informed written consent.

Exclusion Criteria:

* Women who are pregnant or breastfeeding, or planning to become pregnant or breastfeed during the study
* Any sign of active stage III disease as classified by the Centers for Diseases Control and Prevention
* Patients whose antiretroviral therapy contains a strong cytochrome P3A4 inhibitor (ritonavir or cobicistat) or efavirenz
* Patients receiving long-term NSAIDs or corticosteroids
* Patients taking cannabis recreationally
* Patients with a personal history of psychotic disorders
* Patients with a history of severe cerebrovascular disease (ischemic or hemorrhagic stroke)
* Renal failure defined by creatinine clearance <60 mL / min calculated according to MDRD
* Patient with severe hepatic impairment (class C) according to the Child Pugh score
* Unstable liver disease (defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices or persistent jaundice), cirrhosis, known biliary abnormality.
* Disease or history of severe cardiovascular or cerebrovascular disorders (MI, stroke)
* Anticipated need for hepatitis C virus treatment during the randomization phase of the study.
* History or presence of allergy or intolerance to cannabidiol or to the terpenes contained in the study product.
* Active malignant tumor
* Patient who, in the opinion of the investigator, presents a significant risk of suicide
* Any pre-existing physical or mental condition which may interfere with the patient's ability to comply with administration schedules and / or protocol evaluations, or which may compromise patient safety.
* Any condition that is likely to interfere with the absorption, distribution, metabolism, or elimination of study drugs that may prevent the patient from taking oral therapy.
* Non-observant patient
* Persons covered by Article L.1121-5 to L.1121-8 and L.1122-1-2 of the Public Health Code (including minors and protected adults).
* Person under tutorship or curatorship
* Person under safeguard of justice
* Person not affiliated with a social security scheme
* Patient participating in another clinical trial, evaluating a treatment
* Patient with chronic inflammatory disease capable of altering the baseline level of cytokines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Percentage of variation in the quantification of the corresponding mRNAs | Day 0
  Percentage of variation in the quantification of the corresponding mRNAs in the mononuclear cells in the different arms of the study
Percentage of variation in the quantification of the corresponding mRNAs | Week 4
  Percentage of variation in the quantification of the corresponding mRNAs in the mononuclear cells in the different arms of the study
Percentage of variation in the quantification of the corresponding mRNAs | Week 12
  Percentage of variation in the quantification of the corresponding mRNAs in the mononuclear cells in the different arms of the study

SECONDARY OUTCOMES:
Quantifications of the quantities of mRNA in each cell subpopulation | Day 0
  Quantifications of the mRNAs corresponding to S16 and comparison with the data obtained on D0, S4 and S12, and with those obtained from HIV negative donors.
Quantifications of the quantities of mRNA in each cell subpopulation | Week 4
  Quantifications of the mRNAs corresponding to S16 and comparison with the data obtained on D0, S4 and S12, and with those obtained from HIV negative donors.
Quantifications of the quantities of mRNA in each cell subpopulation | Week 12
  Quantifications of the mRNAs corresponding to S16 and comparison with the data obtained on D0, S4 and S12, and with those obtained from HIV negative donors.
Quantification of the Global and targeted methylation (promoters of autophagy genes) of DNA | Day 0
  Quantification of the Global and targeted methylation (promoters of autophagy genes) of DNA and comparison according to the dose administered
Quantification of the Global and targeted methylation (promoters of autophagy genes) of DNA | Week 4
  Quantification of the Global and targeted methylation (promoters of autophagy genes) of DNA and comparison according to the dose administered
Quantification of the Global and targeted methylation (promoters of autophagy genes) of DNA | Week 12
  Quantification of the Global and targeted methylation (promoters of autophagy genes) of DNA and comparison according to the dose administered
Quantification of the mRNAs for autophagy genes and pro and anti-inflammatory cytokines | Day 0
  Quantification of the mRNAs for autophagy genes and pro and anti-inflammatory cytokines and comparison according to the dose administered
Quantification of the mRNAs for autophagy genes and pro and anti-inflammatory cytokines | Week 4
  Quantification of the mRNAs for autophagy genes and pro and anti-inflammatory cytokines and comparison according to the dose administered
Quantification of the mRNAs for autophagy genes and pro and anti-inflammatory cytokines | Week 12
  Quantification of the mRNAs for autophagy genes and pro and anti-inflammatory cytokines and comparison according to the dose administered
Quantification of the dosage of pro and anti-inflammatory cytokines in serum and after in vitro activation of PBMCs | Day 0
  Quantification of the dosage of pro and anti-inflammatory cytokines in serum and after in vitro activation of PBMCs and comparison according to the dose administered
Quantification of the dosage of pro and anti-inflammatory cytokines in serum and after in vitro activation of PBMCs | Week 4
  Quantification of the dosage of pro and anti-inflammatory cytokines in serum and after in vitro activation of PBMCs and comparison according to the dose administered
Quantification of the dosage of pro and anti-inflammatory cytokines in serum and after in vitro activation of PBMCs | Week 12
  Quantification of the dosage of pro and anti-inflammatory cytokines in serum and after in vitro activation of PBMCs and comparison according to the dose administered
Quantification of the expression of the proteins encoded by these same genes | Day 0
  Quantification of the expression of the proteins encoded by these same genes and comparison according to the dose administered
Quantification of the expression of the proteins encoded by these same genes | Week 4
  Quantification of the expression of the proteins encoded by these same genes and comparison according to the dose administered
Quantification of the expression of the proteins encoded by these same genes | Week 12
  Quantification of the expression of the proteins encoded by these same genes and comparison according to the dose administered
Quantification of the autophagic function by detection of positive LC3b vesicles | Day 0
  Quantification of the autophagic function by detection of positive LC3b vesicles and comparison according to the dose administered
Quantification of the autophagic function by detection of positive LC3b vesicles | Week 4
  Quantification of the autophagic function by detection of positive LC3b vesicles and comparison according to the dose administered
Quantification of the autophagic function by detection of positive LC3b vesicles | Week 12
  Quantification of the autophagic function by detection of positive LC3b vesicles and comparison according to the dose administered
Quantification of the activation (CD38, HLA-DR) and degree of senescence (CD57, PD1) of CD4 and CD8 lymphocytes and monocytes (CD16, HLA-DR) | Day 0
  Quantification of the activation (CD38, HLA-DR) and degree of senescence (CD57, PD1) of CD4 and CD8 lymphocytes and monocytes (CD16, HLA-DR) and comparison according to the dose administered
Quantification of the activation (CD38, HLA-DR) and degree of senescence (CD57, PD1) of CD4 and CD8 lymphocytes and monocytes (CD16, HLA-DR) | Week 4
  Quantification of the activation (CD38, HLA-DR) and degree of senescence (CD57, PD1) of CD4 and CD8 lymphocytes and monocytes (CD16, HLA-DR) and comparison according to the dose administered
Quantification of the activation (CD38, HLA-DR) and degree of senescence (CD57, PD1) of CD4 and CD8 lymphocytes and monocytes (CD16, HLA-DR) | Week 12
  Quantification of the activation (CD38, HLA-DR) and degree of senescence (CD57, PD1) of CD4 and CD8 lymphocytes and monocytes (CD16, HLA-DR) and comparison according to the dose administered
Quantification of T3, T4, T8, NK, NK-T, B populations, monocytes. | Day 0
  Quantification of T3, T4, T8, NK, NK-T, B populations, monocytes and comparison according to the dose administered
Quantification of T3, T4, T8, NK, NK-T, B populations, monocytes. | Week 4
  Quantification of T3, T4, T8, NK, NK-T, B populations, monocytes and comparison according to the dose administered
Quantification of T3, T4, T8, NK, NK-T, B populations, monocytes. | Week 12
  Quantification of T3, T4, T8, NK, NK-T, B populations, monocytes and comparison according to the dose administered
Measurement of DNA-HIV in PBMCs | Day 0
Measurement of DNA-HIV in PBMCs | Week 4
Measurement of DNA-HIV in PBMCs | Week 12
Incidence and severity of AEs and laboratory abnormalities | Week 12
Proportion of patients who discontinued treatment due to AE | Week 12
Determination of CBD in the blood at W12, compared to assays S0 and S16 | Week 12
Quality of life questionnaire | Day 0
  It is a self-assessment quality of life scale comprising 11 questions
Quality of life questionnaire | Week 4
  It is a self-assessment quality of life scale comprising 11 questions
Quality of life questionnaire | Week 12
  It is a self-assessment quality of life scale comprising 11 questions

CONTACTS AND LOCATIONS:
Overall Officials: Thierry PRAZUCK, Dr, Principal Investigator — CHR d'Orléans
Locations (1):
- Centre Hospitalier Régional d'Orléans, France, Orléans, France

REFERENCES:
- [Background] Guittaut M, Charpentier S, Normand T, Dubois M, Raimond J, Legrand A. Identification of an internal gene to the human Galectin-3 gene with two different overlapping reading frames that do not encode Galectin-3. J Biol Chem. 2001 Jan 26;276(4):2652-7. doi: 10.1074/jbc.m002523200. PMID 11160123
- [Background] Raimond J, Rouleux F, Monsigny M, Legrand A. The second intron of the human galectin-3 gene has a strong promoter activity down-regulated by p53. FEBS Lett. 1995 Apr 17;363(1-2):165-9. doi: 10.1016/0014-5793(95)00310-6. PMID 7729540
- [Background] Gonzalez P, Robinet P, Charpentier S, Mollet L, Normand T, Dubois M, Legrand A. Apoptotic activity of a nuclear form of mitogaligin, a cell death protein. Biochem Biophys Res Commun. 2009 Jan 23;378(4):816-20. doi: 10.1016/j.bbrc.2008.11.133. Epub 2008 Dec 9. PMID 19071086
- [Background] Duneau M, Boyer-Guittaut M, Gonzalez P, Charpentier S, Normand T, Dubois M, Raimond J, Legrand A. Galig, a novel cell death gene that encodes a mitochondrial protein promoting cytochrome c release. Exp Cell Res. 2005 Jan 15;302(2):194-205. doi: 10.1016/j.yexcr.2004.08.041. PMID 15561101
- [Background] Robinet P, Mollet L, Gonzalez P, Normand T, Charpentier S, Brule F, Dubois M, Legrand A. The mitogaligin protein is addressed to the nucleus via a non-classical localization signal. Biochem Biophys Res Commun. 2010 Jan 29;392(1):53-7. doi: 10.1016/j.bbrc.2009.12.162. Epub 2010 Jan 7. PMID 20056110